CLINICAL TRIAL: NCT05002855
Title: Effect of Implementation of Enhanced Recovery After Surgery (ERAS) Protocol on 3-year Survival After Colorectal Surgery for Cancer - a Retrospective Cohort of 1001 Patients
Brief Title: Effect of Implementation of Enhanced Recovery After Surgery on 3-year Survival After Colorectal Surgery for Cancer
Acronym: RACCOR
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2021
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Enhanced Recovery After Surgery (ERAS)
  Interventions: Other: Enhanced Recovery After Surgery (ERAS)
- Conventional Recovery Strategy (pre-ERAS)

INTERVENTIONS:
Other: Enhanced Recovery After Surgery (ERAS) — Multidisciplinary approach to perioperative care.
  Groups: Enhanced Recovery After Surgery (ERAS)

SUMMARY:
Several recent studies have shown that the Enhanced Recovery After Surgery (ERAS) protocol reduces morbidity and mortality and shortens the length of stay compared to conventional recovery strategy (pre-ERAS). The aim of this study was to evaluate the effect of the implementation of this protocol on 3-year overall survival and postoperative outcome in patients undergoing colorectal resection for cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aadult patients, who had undergone resection for colorectal cancer or a precancerous lesion and were cared for using the ERAS protocol or received conventional care (pre-ERAS).
* Informed patients

Exclusion Criteria:

* Patients presenting or developing peritoneal cancer,
* Patients having resection for palliative reasons,
* Patients those under curatorship or tutelage
* Opposed patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consisted of all consecutive adult patients, who had undergone resection for colorectal cancer or a precancerous lesion and were cared for using the ERAS protocol or received conventional care (pre-ERAS). The records of consecutive patients recorded in the hospital's electronic medical records (PMSI) between January 2005 and December 2017 were screened. Non-inclusion criteria included patients presenting or developing peritoneal cancer, patients having resection for palliative reasons, those under curatorship or tutelage.
Sampling Method: Non-Probability Sample
Enrollment: 1001 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of the implementation of this protocol on 3-year overall survival. | 3 years
  3-year overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Faucheron, Study Director — CHU Grenoble Alpes
Locations (1):
- Jean-Luc Faucheron, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alfonsi P, Slim K, Chauvin M, Mariani P, Faucheron JL, Fletcher D; le groupe de travail de la Societe francaise d'anesthesie et reanimation (Sfar) et de la Societe francaise de chirurgie digestive (SFCD). [Guidelines for enhanced recovery after elective colorectal surgery]. Ann Fr Anesth Reanim. 2014 May;33(5):370-84. doi: 10.1016/j.annfar.2014.03.007. Epub 2014 May 20. French. PMID 24854967
- [Result] Gignoux B, Gosgnach M, Lanz T, Vulliez A, Blanchet MC, Frering V, Faucheron JL, Chasserant P. Short-term Outcomes of Ambulatory Colectomy for 157 Consecutive Patients. Ann Surg. 2019 Aug;270(2):317-321. doi: 10.1097/SLA.0000000000002800. PMID 29727328
- [Result] Faucheron JL, Trilling B, Sage PY. Ambulatory colectomy: fast-track management pushed to its limits? Tech Coloproctol. 2018 Oct;22(10):741-742. doi: 10.1007/s10151-018-1871-5. Epub 2018 Nov 9. No abstract available. PMID 30413997
- [Result] Trilling B, Sage PY, Faucheron JL. What is fast track multimodal management of colorectal cancer surgery in real life? Tech Coloproctol. 2018 May;22(5):401-402. doi: 10.1007/s10151-018-1799-9. Epub 2018 Jun 1. No abstract available. PMID 29855815
- [Result] Carrier G, Cotte E, Beyer-Berjot L, Faucheron JL, Joris J, Slim K; Groupe Francophone de Rehabilitation Amelioree apres Chirurgie (GRACE). Post-discharge follow-up using text messaging within an enhanced recovery program after colorectal surgery. J Visc Surg. 2016 Aug;153(4):249-52. doi: 10.1016/j.jviscsurg.2016.05.016. Epub 2016 Aug 8. PMID 27423211
- [Result] Slim K, Delaunay L, Joris J, Leonard D, Raspado O, Chambrier C, Ostermann S; Le Groupe francophone de rehabilitation amelioree apres chirurgie (GRACE). How to implement an enhanced recovery program? Proposals from the Francophone Group for enhanced recovery after surgery (GRACE). J Visc Surg. 2016 Dec;153(6S):S45-S49. doi: 10.1016/j.jviscsurg.2016.05.008. Epub 2016 Jun 14. No abstract available. PMID 27316295
- [Result] Faujour V, Slim K, Corond P. [The future, in France, of enhanced recovery after surgery seen from the economical perspective]. Presse Med. 2015 Jan;44(1):e23-31. doi: 10.1016/j.lpm.2014.07.021. Epub 2014 Dec 22. French. PMID 25540876
- [Result] Launay-Savary MV, Mathonnet M, Theissen A, Ostermann S, Raynaud-Simon A, Slim K; GRACE (Groupe francophone de Rehabilitation Amelioree apres Chirurgie). Are enhanced recovery programs in colorectal surgery feasible and useful in the elderly? A systematic review of the literature. J Visc Surg. 2017 Feb;154(1):29-35. doi: 10.1016/j.jviscsurg.2016.09.016. Epub 2016 Nov 11. PMID 27842907